CLINICAL TRIAL: NCT04134832
Title: Clinicopathological Assessment of Pancreatic Neuroendocrine Tumors and Carcinomas in Alsace Region
Brief Title: Study of Pancreatic Neuroendocrine Tumors and Carcinomas in Alsace Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7435
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Neuroendocrine Tumor
Keywords: Pancreatic neuroendocrine tumors; Neutrophil-to-lymphocyte ratio
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic Neuroendocrine tumors and carcinomas (pNET) see the last year their incidence and prevalence going up. On the basis of their grade of differentiation and proliferation ratio measured Ki67 staining, there are divided into 3 grade groups : Grade 1 with Ki67 between 1 and 3%, Grade 2 between 3 and 20% and well-differentiated neuroendocrine grade tumors 3 with KI67 greater than 20%, so undifferentiated carcinomas.

pNET is a heterogenous group of tumors with variable prognosis. The aim of this study is to identify the prognostic factors in this population, as well the place of neutrophil-to-lymphocyte ratio as a prognostic marker. The primary endpoint is the description of clinic and pathological parameters of patients from Alsace. The secondary endpoints are the identification of prognostic factors in this population

ELIGIBILITY:
Inclusion criteria:

1. Major topic ((≥18 years)
2. Subject with histologically confirmed pancreatic neuroendocrine tumor or carcinoma
3. Subject with tumours or neuroendocrine carcinoma of the pancreas at any stage of the disease.
4. Subject covered in one of the participating centres between 01/01/2008 and 01/01/2019
5. Have a pre-therapeutic biological check-up
6. Subject who has not expressed opposition to the use of his or her data for research purposes

Exclusion criteria:

1. Subject who expressed opposition to participate in the study
2. Lack of histological data
3. Minor subject
4. Patient under the protection of justice
5. Subject under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with histologically confirmed pancreatic neuroendocrine tumor or carcinoma, with tumours or neuroendocrine carcinoma of the pancreas at any stage of the disease and covered in one of the participating centres between 01/01/2008 and 01/01/2019
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The survival will be evaluated by Kaplan Meier Method. The prognostic factors will be evaluated with univariate and multivariate analysis by Cox regression model. | The participant will be followed-up for a maximum of 11 years, and 1 year at least.

CONTACTS AND LOCATIONS:
Locations (1):
- Service D'Hematologie Et D'Oncologie, Strasbourg, France